CLINICAL TRIAL: NCT07342933
Title: Outcomes of Children in Whom a Prenatal Exome Was Performed Based on Ultrasound Findings
Acronym: ExoPré
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9815
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Amniocentesis Affecting Fetus
Keywords: Amniocentesis Affecting Fetus; Prenatal Exome; Ultrasound Findings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amniocentesis is a test offered to couples based on ultrasound findings during pregnancy. Currently, genetic analysis using FISH and ACPA is routinely performed. For the past four years, additional exome sequencing has been offered after two ultrasound findings, if FISH and ACPA are negative. In this study, investigators aim to review the results of this exome sequencing analysis, examine the outcomes obtained, and study the outcomes of the children after birth. Can parents be completely reassured when the exome sequencing is negative, or does this indicate that investigators are not yet sufficiently sensitive in their genetic analysis?

ELIGIBILITY:
Inclusion Criteria:

* Child under 4 years of age
* Exome sequencing performed at the Strasbourg University Hospitals (HUS) following amniocentesis during pregnancy between November 2021 and September 2025.

Exclusion Criteria:

* Refusal to participate in the study
* Exome sequencing not performed at the Strasbourg University Hospital.
* Lack of prenatal ultrasound information.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child under 4 years of age having an exome sequencing performed at the Strasbourg University Hospitals following amniocentesis during pregnancy between November 2021 and September 2025.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Psychomotor development of the children | Up to 24 months
  Psychomotor development of the children based on items from the health record:
  The items in the child's health record are used to:
  * monitor the child's normal development,
  * detect any potential delays early, and
  * reassure parents or refer them to a professional if needed.
  Example: If a child is not yet walking at 18 months:
  * this is not necessarily serious,
  * but it may lead the doctor to suggest monitoring or exercises.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologique et d'Obstétrique - CHU de Strasbourg - France, Strasbourg, France